CLINICAL TRIAL: NCT03161171
Title: Behavioral Challenges in Children With Mucopolysaccharidosis Type I-III and Parental Coping Strategies
Brief Title: Parental Coping With Challenging Behavior in Mucopolysaccharidosis Type I-III
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Markus Ries, MD PhD MHSc FCP, Professor, University Hospital Heidelberg
Other Study IDs: 01
Record Dates: First submitted 2017-04-24; First posted 2017-05-19 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Mucopolysaccharidosis Type I; Mucopolysaccharidosis Type II; Mucopolysaccharidosis Type III; Behavior Disorders; Coping Behavior
MeSH Terms: conditions — Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis III; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is an observational study — This is an observational study

SUMMARY:
The study quantitates behavioral challenges in mucopolysaccharidosis type I-III and parental coping strategies

DETAILED DESCRIPTION:
This is a prospective, cross-sectional, observational study quantitatively assessing

1. challenging behavior in children with MPS, an orphan, progressive, neurodegenerative metabolic disorder, and
2. parental coping strategies for this challenging behavior.

Patients registered at the German Society for Mucopolysacchardoses giving written informed consent are eligible. The study is based on questionnaires. IRB approval was obtained.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mucopolysaccharidosis type I, II or III
* Written informed consent
* Patient is registered at the German Society for Mucopolysaccharidosis

Exclusion Criteria:

* Patient / Family does not give written informed consent.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with mucopolysaccharidosis type I-III below 18 years of age registered at the German Society for Mucopolysaccharidosis
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
Coping strategies for challenging behavior and for family burden in mucopolysaccharidosis type I-III | 10 minutes
  assessed by visual analogue scale

SECONDARY OUTCOMES:
Quantity of behavioral abnormalities in children with mucopolysaccharidosis type I-III | 10 minutes
  assessed by visual analogue scale
Intensity of behavioral abnormalities in children with mucopolysaccharidosis type I-III | 10 minutes
  assessed by visual analogue scale
Psychosocial burden in families with mucopolysaccharidosis type I-III | 10 minutes
  assessed by visual analogue scale
Psychosocial burden in families with mucopolysaccharidosis type I-III | 10 minutes
  assessed by Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Markus Ries, MD PhD MHSc FCP, Principal Investigator — markus.ries@med.uni-heidelberg.de
Locations (1):
- University of Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoffmann F, Hoffmann S, Kunzmann K, Ries M. Challenging behavior in mucopolysaccharidoses types I-III and day-to-day coping strategies: a cross sectional explorative study. Orphanet J Rare Dis. 2020 Oct 2;15(1):275. doi: 10.1186/s13023-020-01548-9. PMID 33008435